CLINICAL TRIAL: NCT01268254
Title: The Red Wine Project: a Study of Ageing Indexes and Prevalence of Atherosclerosis in Regular Red Wine Consumers Versus Abstainers
Brief Title: Red Wine and Ageing and Atherosclerosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Protasio Lemos da Luz/ Cardiology Professor, Heart Insitute (InCor) Clinical Hospital of School Medicine University of Sao Paulo
Other Study IDs: 1-48200805
Record Dates: First submitted 2010-12-28; First posted 2010-12-29 (Estimated); Last update posted 2010-12-29 (Estimated); Status verified 2010-09

CONDITIONS: Coronary Disease
Keywords: wine; aging; atherosclerosis; telomere; tomography; coronary vessels
MeSH Terms: conditions — Coronary Disease; Atherosclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — total blood sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- red wine: red wine usual consumer versus abstemious

SUMMARY:
The investigators will evaluate 100 regular red wine consumer men and 100 abstainers men from 50 years-old to 70 years-old by coronary risk prevalence, mood status, anthropometric measures, daily caloric ingest, lipid profile, carotid intimal media thickness, brachial flow mediate dilatation, coronary tomographic angiography and leucocyte telomere length.

The sample size has been calculated expecting that regular red wine ingestion would lead to a five year old younger vascular ageing indexes measured by carotid intimal media thickness, coronary artery calcium scores and leucocyte telomere length longer than those abstainers subjects at same age.

The investigators hypothesized that regular wine consumers present less coronary lesion and coronary calcium score on coronary tomographic angiography, lower carotid intimal media thickness and higher mean telomere length due the benefice of wine.

ELIGIBILITY:
Inclusion Criteria:

* healthy male, from 50 years-old to 70 years-old.

Exclusion Criteria:

* asiatic or with manifest atherosclerosis disease

Ages: 50 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: male subjects, between 50 years-old and 70 years-old, divided in 2 groups: usual red wine consumers and red wine abstemious
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2009-10; Primary Completion 2011-03 (Estimated); Study Completion 2011-04 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Protasio L Da Luz, MD, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Heart Insitute ( InCor) University of Sao Paulo, São Paulo, São Paulo, Brazil